CLINICAL TRIAL: NCT06611410
Title: 1 Week Crossover Dispensing Study: Buttermere Versus MiSight 1 Day Soft Contact Lenses
Brief Title: 1 Week Crossover Study Between Two Soft Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CV-23-59
Record Dates: First submitted 2024-09-23; First posted 2024-09-25 (Actual); Results first posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-08

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Test Lenses, Then Control Lenses (Experimental): Participants will wear the Test Lenses in both eyes for one week and then cross over to the Control Lenses in both eyes for one week.
  Interventions: Device: Test Lenses (stenfilcon A); Device: Control Lenses (omafilcon A)
- Control Lenses, Then Test Lenses (Experimental): Participants will wear the Control Lenses in both eyes for one week and then cross over to the Test Lenses in both eyes for one week.
  Interventions: Device: Test Lenses (stenfilcon A); Device: Control Lenses (omafilcon A)

INTERVENTIONS:
Device: Test Lenses (stenfilcon A) — Daily disposable, soft contact lenses worn for one week.
Device: Control Lenses (omafilcon A) — Daily disposable, soft contact lenses worn for one week.

SUMMARY:
The objective of this investigation is to compare the visual clinical performance of two daily disposable soft contact lenses.

DETAILED DESCRIPTION:
This is a prospective, multiple day, double (investigator and subject) masked, randomized, bilateral crossover study comparing a Test lens against an appropriate Control lens. Main aim is to compare visual acuity and subjective vision ratings of vision quality between two lenses in habitual soft lens wearers.

ELIGIBILITY:
Inclusion Criteria:

* Are 8 to 18 years of age (inclusively)
* Have read, signed and dated:

  * Age 18 - The Participant Informed Consent Form (participant only)
  * Age 12-17 - The Parental Permission Form (participant and parent)
  * Age 8-11 - The Parental Permission Form (parent) and Assent form (participant)
* Are willing and able to follow instructions and maintain the appointment schedule.
* Are habitual daily wearers of spherical single vision soft contact lenses to correct for distance vision in each eye, including myopia control soft contact lenses as below-
* Currently wears spherical soft contact lenses or myopia control soft contact lenses.
* Have a pair of wearable back-up spectacles.
* Are willing and able to wear contact lenses for at least 10 hours a day, 6 days a week while in the study.
* Are myopic with subjective refraction: -0.75D to -7.00D spherical, with an astigmatism ≤ -0.75D in each eye with maximum spherical equivalent anisometropia of 1.00D
* Are correctable to a visual acuity of +0.10 logMAR or better (in each eye) with sphero-cylindrical subjective refraction.
* Have clear corneas with no corneal scars or any active ocular disease.
* Can be fit with the study contact lenses with a power between -0.75 and -7.00 DS; this translates to best corrected vision sphere refraction that vertexes to a CL power between -0.75 and -7.00 (inclusive) at screening visit.
* Demonstrate an acceptable fit with the study contact lenses.
* Demonstrate that they can safely and independently insert and remove contact lenses at the screening/fitting visit.

Exclusion Criteria:

* Have taken part in another clinical research study within the last 14 days.
* Are currently habitual wearers of toric contact lenses.
* Have worn any rigid contact lenses or ortho-keratology contact lenses in the past 30 days.
* Are an extended contact lens wearer (i.e., sleeping with their contact lenses).
* Are on ongoing atropine treatment for myopia control.
* Have a difference of > 1.0 D in best vision sphere subjective refraction between eyes.
* Have amblyopia and/or strabismus/binocular vision problem.
* Have any known active ocular disease, allergies and/or infection.
* Have a systemic condition that in the opinion of the investigator may affect a study outcome variable.
* Are using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable.
* Have a known sensitivity to the diagnostic pharmaceuticals to be used in the study.
* Have undergone refractive error surgery or intraocular surgery.
* Are a member of CORL directly involved in the study.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2024-06-05 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pete S Kollbaum, OD, PhD, Principal Investigator — Indiana University
Locations (1):
- Clinical Optics Research Lab (CORL), Bloomington, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Ten participants were enrolled in the study. One participant was excluded due to screening failure. (n=9)
Groups:
- Test Lenses First, Then Control Lenses: Participants wore the Test Lenses in both eyes for one week and then crossed over to the Control Lenses in both eyes for one week.
- Control Lenses First, Then Test Lenses: Participants wore the Control Lenses in both eyes for one week and then crossed over to the Test Lenses in both eyes for one week.
Period: (Period 1): First Intervention (7 Days)
Arm/Group | Test Lenses First, Then Control Lenses | Control Lenses First, Then Test Lenses
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0
Period: (Period 2): Second Intervention (7 Days)
Arm/Group | Test Lenses First, Then Control Lenses | Control Lenses First, Then Test Lenses
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Total eight participants were analyzed who completed all study visits. (One participant was excluded from the analysis due to protocol deviation)
Arm/Group | Overall Study
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: High Contrast, Binocular, Distance Visual Acuity (logMAR)
Description: High contrast, binocular, distance visual acuity (logMAR) will be measured at 1-week visit.
Time Frame: At the end of one week wear
Population: Analysis population includes all the participants who completed all the study visits.
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- Test Lenses (Stenfilcon A): Participants that received the Test Lenses and completed all study visits
- Control Lenses (Omafilcon A): Participants that received the Control Lenses and completed all study visits
Arm/Group | Test Lenses (Stenfilcon A) | Control Lenses (Omafilcon A)
Number analyzed (Participants) | 8 | 8
logMAR | -0.15 (0.03) | -0.15 (0.05)

2. Secondary Outcome: Subjective Vision Quality
Description: Subjective vision quality on 0-100 Visual Analog Scale (where, 0=very poor and 100=very good)
Time Frame: At the end of one week wear
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Lenses (Stenfilcon A) | Control Lenses (Omafilcon A)
Number analyzed (Participants) | 8 | 8
units on a scale | 94.12 (4.67) | 87.12 (11.61)

ADVERSE EVENTS:
Time Frame: Duration study, approximately 20 days.
Groups:
- Test Lenses (Stenfilcon A): All participants that received the Test Lenses
- Control Lenses (Omafilcon A): All participants that received the Control Lenses
Arm/Group | Test Lenses (Stenfilcon A) | Control Lenses (Omafilcon A)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 1/9 | 1/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Lenses (Stenfilcon A) (N=9) | Control Lenses (Omafilcon A) (N=9)
Viral Conjuctivitis (Eye disorders) | 1 (1) | 0 (0)
Lightheaded (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-07): https://cdn.clinicaltrials.gov/large-docs/10/NCT06611410/Prot_SAP_000.pdf